CLINICAL TRIAL: NCT04379518
Title: Phase 1/2A Study of Rintatolimod and IFN Alpha Regimen in Cancer Patients With COVID-19
Brief Title: Rintatolimod and IFN Alpha-2b for the Treatment of COVID-19 in Cancer Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AIM ImmunoTech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 659920; NCI-2020-02317 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 659920 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2020-05-06; First posted 2020-05-07 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Symptomatic COVID-19 Infection Laboratory-Confirmed
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Introns; Interferon alpha-2; poly(I).poly(c12,U)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Rintatolimod, recombinant interferon alfa-2b 0 MU/M^2 (Experimental): Dose level 1:Patients receive rintatolimod IV over 2.5-3 hours plus recombinant interferon alfa-2b IV 0 over 20 minutes on day 1 and on day 3 (or 4) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Recombinant Interferon Alfa-2b; Drug: Rintatolimod
- Rintatolimod, recombinant interferon alfa-2b 5 MU/M^2 (Experimental): Dose level 2 :Patients receive rintatolimod IV over 2.5-3 hours plus recombinant interferon alfa-2b IV 5 MU/M^2 over 20 minutes on day 1 and on day 3 (or 4) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Recombinant Interferon Alfa-2b; Drug: Rintatolimod
- Rrintatolimod plus Standard of Care) (Experimental): Patients receive rintatolimod IV over 2.5-3 hours once plus standard of care.
  Interventions: Drug: Rintatolimod
- Rintatolimod, recombinant interferon alfa-2b 10 MU/M^2 (Experimental): Dose level 3: Patients receive rintatolimod IV over 2.5-3 hours plus recombinant interferon alfa-2b IV 10 MU/M^2 over 20 minutes on day 1 and on day 3 (or 4) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Recombinant Interferon Alfa-2b; Drug: Rintatolimod
- Rintatolimod, recombinant interferon alfa-2b 20 MU/M^2 (Experimental): Dose level 4: Patients receive rintatolimod IV over 2.5-3 hours plus recombinant interferon alfa-2b IV 20 MU/M^2 over 20 minutes on day 1 and on day 3 (or 4) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Recombinant Interferon Alfa-2b; Drug: Rintatolimod

INTERVENTIONS:
Biological: Recombinant Interferon Alfa-2b — Given IV
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; Interferon alfa 2b; Interferon Alfa-2B; Interferon Alpha-2b; Intron A; Sch 30500; Urifron; Viraferon
  Arms: Rintatolimod, recombinant interferon alfa-2b 0 MU/M^2; Rintatolimod, recombinant interferon alfa-2b 10 MU/M^2; Rintatolimod, recombinant interferon alfa-2b 20 MU/M^2; Rintatolimod, recombinant interferon alfa-2b 5 MU/M^2
Drug: Rintatolimod — Given IV
  Other Names: Ampligen; Atvogen

SUMMARY:
This phase I/IIa trial studies the best dose and side effects of rintatolimod and interferon (IFN) alpha-2b in treating cancer patients with COVID-19 infection. Interferon alpha is a protein important for defense against viruses. It activates immune responses that help to clear viral infection. Rintatolimod is double stranded ribonucleic acid (RNA) designed to mimic viral infection by stimulating immune pathways that are normally activated during viral infection. Giving rintatolimod and interferon alpha-2b may activate the immune system to limit the replication and spread of the virus.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of the combination of intravenous (i.v.) rintatolimod administered with or without i.v. IFN alpha (recombinant interferon alfa-2b [Intron A]) in patients with cancer with coronavirus disease 2019 (COVID-19).

II. Determine the kinetics of viral load in nasopharyngeal swabs in the course of treatment and Days 7 and 14.

SECONDARY OBJECTIVES:

I. To assess the efficacy of the treatment combination in patients with cancer with COVID-19.

II. Determine the kinetics of viral load in the peripheral blood in the course of treatment and Days 7 and 14.

III. Determine the kinetics of changes of the immune subsets and circulating inflammatory mediators (including C-reactive protein [CRP], cytokines, chemokines, interferons) in peripheral blood in the course of treatment and Days 7 and 14.

IV. Determine the induction of known mediators of antiviral immunity that include (myxovirus resistance gene, MxA; protein Kinase R (PKR); oligoadenylate synthetase-2 (OAS2); RNAse-L, IFN-stimulated gene-15 (ISG15); IFN-induced proteins with tetratricopeptide repeats (IFIT1) and IFN-inducible transmembrane protein 3 (IFITM3), TLR3, RIG-I, MDA5, IRF3, IRF7, in nasopharyngeal swabs material and blood cells of patients on all tiers of treatment.

OUTLINE: This is a phase I, dose-escalation study of recombinant interferon alfa-2b followed by a phase II study.

LEAD-IN PHASE: Patients receive rintatolimod IV over 2.5-3 hours on day 1 and day 3 (or 4).

ARM I: Patients receive rintatolimod IV over 2.5-3 hours and recombinant interferon alfa-2b IV over 20 minutes on day 1 and on day 3 or 4 in the absence of disease progression or unacceptable toxicity.

EXPANSION COHORT:

ARM III: Patients receive rintatolimod IV over 2.5-3 hours along with standard of care.

Patients are followed up at days 7, 14 and 30 after initiation of the study regimen.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA (MAIN COHORT):
* Patients with cancer, with the exception of patients with active acute leukemia and allogeneic hematopoietic stem cell transplant recipients. Patients may be on active therapy or received therapy (e.g., chemotherapy, radiation or surgery) within 7 years. Patients with active cancer who have not yet been treated (e.g. newly diagnosed cancer or early stage myelodysplastic syndrome [MDS] or chronic lymphocytic leukemia [CLL]) are eligible. Basal cell cancer and carcinoma in situ treated with local excision alone do not qualify for inclusion
* Presence of symptomatic infection, defined by fever (temperature [T] >= 38 degrees Celsius [C]) OR respiratory symptoms (cough, nasal congestion, or shortness of breath) OR lung infilitrates on chest X-ray or CT imaging. Diagnosis of COVID-19 is based on polymerase chain reaction (PCR) testing of respiratory samples.
* Age equal to >= 18 years or older (children are excluded because COVID-19 typically has a milder course in children, and lack of safety data of this regimen in children)
* Platelet >= 75,000/uL
* Hemoglobin >= 9 g/dL
* Hematocrit >= 27%
* Absolute neutrophil count (ANC) >= 1000/uL
* Creatinine clearance >= 50 mL/min (Cockcroft-Gault Equation-note: plasma creatine instead of serum is used at Roswell Park)
* Total bilirubin =< 2 X institutional upper limit of normal (ULN)
* Aspartate transaminase (AST) (plasma) and alanine transferase (ALT) (plasma) =< 2 X institutional ULN
* Plasma amylase and lipase =< 2 X institutional ULN
* In the absence of COVID-19, a life expectancy of 6 months is expected
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* NOTE: For blood chemistry labs, Roswell Park clinical blood chemistries are performed on plasma unless otherwise indicated
* EXPANSION COHORT: Patients with cancer or allogeneic stem cell transplant recipients with and without a cancer diagnosis

  * Patients with cancer may be on active therapy or received therapy (e.g., chemotherapy, radiation or surgery) within 7 years
  * Patients with active cancer who have not yet been treated (e.g. newly diagnosed cancer or early stage MDS or CLL) are eligible
  * Basal cell cancer and carcinoma in situ treated with local excision alone do not qualify for inclusion
* Presence of symptomatic infection, defined by fever (T >= 38.0 degrees C ) OR respiratory symptoms (cough, nasal congestion, or shortness of breath) OR lung infiltrates by chest X-ray or CT imaging. Diagnosis of COVID-19 is based on PCR testing of respiratory samples. Severe infection is excluded
* Age equal to >= 18 years or older (children are excluded because COVID-19 typically has a milder course in children, and lack of safety data of this regimen in children). In the absence of COVID-19, a life expectancy of 6 months is expected
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure. There may be specific instances when the patient can't provide informed consent, e.g. they require mechanical ventilation and are sedated, in which case a health care proxy will be able to provide informed consent. Patients with temporary cognitive impairment will be consented once their capacity has returned. Patients with chronic cognitive impairment, e.g. dementia, that precludes informed consent will not be enrolled.

Exclusion Criteria:

* EXCLUSION CRITERIA (MAIN COHORT):
* Patients with severe COVID-19 infection defined by pulmonary infiltrates on chest x-ray or computed tomography (CT) imaging plus one of the following: room air oxygen saturation (SaO2) =< 92%, room air partial pressure of oxygen (PaO2) < 70 mm Hg, or partial pressure of oxygen in arterial blood (PaO2)-PaO2 (alveolar gas) >= 35 mm Hg
* Contraindication to recombinant (r)-INFalpha based on prior hypersensitivity, autoimmune hepatitis, decompensated liver disease
* Patients who have active acute myeloid leukemia or acute lymphoid leukemia or are allogeneic hematopoietic stem transplant recipients. Acute leukemia in remission and chronic leukemias are not exclusion criteria
* Cardiac events:

  * Acute coronary syndrome, myocardial infarction, or ischemia within past 3 months
  * New York Heart Association classification of III or IV congestive heart failure
* Unwilling or unable to follow protocol requirements
* Patients with known serious mood disorders
* Any additional condition, such as pre-existing inflammatory lung disease, which in the investigator's opinion deems the participant an unsuitable candidate to receive the study drugs
* Concurrent infections, e.g. bacterial pneumonia or sepsis, that would make it difficult to evaluate clinical response to therapy or study drug toxicities
* Therapies known to cause cytokine release syndrome (CRS), e.g. engineered T cells, within 30 days
* Patients at high risk for tumor lysis syndrome
* Concurrent active pneumonitis predating COVID-19, such as from checkpoint inhibitor therapy, chemotherapy-associated toxicity, or radiation pneumonitis
* Autoimmune disease that requires systemic immunosuppression
* Protocol-defined baseline abnormalities in cell counts, renal, or hepatic function
* Any additional condition which in the investigator's opinion deems the participant an unsuitable candidate to receive the study drugs
* EXCLUSION CRITERIA: EXPANSION COHORT:
* Patients with respiratory failure requiring mechanical ventilation with FIO2 of > 60%.
* Allogeneic hematopoietic stem cell transplant recipients with active pulmonary graft versus host disease (GvHD) (any grade)
* Cardiac events:

  * Acute coronary syndrome, myocardial infarction, or ischemia within past 3 months,
  * New York Heart Association classification of III or IV congestive heart failure
* Unwilling or unable to follow protocol requirements
* Any additional condition which in the investigator's opinion deems the participant an unsuitable candidate to receive the study drugs
* Cognitively impaired adults/adults with impaired decision-making capacity
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igor Puzanov, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2: Dose level 1:Patients receive rintatolimod IV over 2.5-3 hours plus recombinant interferon alfa-2b IV 0 over 20 minutes on day 1 and on day 3 (or 4) in the absence of disease progression or unacceptable toxicity.
  Biological/Vaccine: Recombinant Interferon Alfa-2b Given IV
  Other Names:
  Alfatronol Glucoferon Heberon Alfa IFN alpha-2B Interferon alfa 2b Interferon Alfa-2B Interferon Alpha-2b Intron A recombinant interferon alfa-2b Sch 30500 Urifron Viraferon Drug: Rintatolimod Given IV
  Other Names:
  Ampligen Atvogen RINTATOLIMOD
- 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2: Dose level 2 :Patients receive rintatolimod IV over 2.5-3 hours plus recombinant interferon alfa-2b IV 5 MU/M^2 over 20 minutes on day 1 and on day 3 (or 4) in the absence of disease progression or unacceptable toxicity.
  Biological/Vaccine: Recombinant Interferon Alfa-2b Given IV
  Other Names:
  Alfatronol Glucoferon Heberon Alfa IFN alpha-2B Interferon alfa 2b Interferon Alfa-2B Interferon Alpha-2b Intron A recombinant interferon alfa-2b Sch 30500 Urifron Viraferon Drug: Rintatolimod Given IV
  Other Names:
  Ampligen Atvogen RINTATOLIMOD
- 3. Experimental: Rrintatolimod Plus Standard of Care): Patients receive rintatolimod IV over 2.5-3 hours once plus standard of care.
  Drug: Rintatolimod Given IV
  Other Names:
  Ampligen Atvogen RINTATOLIMOD
- 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2: Dose level 3: Patients receive rintatolimod IV over 2.5-3 hours plus recombinant interferon alfa-2b IV 10 MU/M^2 over 20 minutes on day 1 and on day 3 (or 4) in the absence of disease progression or unacceptable toxicity.
  Biological/Vaccine: Recombinant Interferon Alfa-2b Given IV
  Other Names:
  Alfatronol Glucoferon Heberon Alfa IFN alpha-2B Interferon alfa 2b Interferon Alfa-2B Interferon Alpha-2b Intron A recombinant interferon alfa-2b Sch 30500 Urifron Viraferon Drug: Rintatolimod Given IV
  Other Names:
  Ampligen Atvogen RINTATOLIMOD
- 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2: Dose level 4: Patients receive rintatolimod IV over 2.5-3 hours plus recombinant interferon alfa-2b IV 20 MU/M^2 over 20 minutes on day 1 and on day 3 (or 4) in the absence of disease progression or unacceptable toxicity.
  Biological/Vaccine: Recombinant Interferon Alfa-2b Given IV
  Other Names:
  Alfatronol Glucoferon Heberon Alfa IFN alpha-2B Interferon alfa 2b Interferon Alfa-2B Interferon Alpha-2b Intron A recombinant interferon alfa-2b Sch 30500 Urifron Viraferon Drug: Rintatolimod Given IV
  Other Names:
  Ampligen Atvogen RINTATOLIMOD
Period: Overall Study
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Started | 4 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2 | Total
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (6.0) |  |  |  |  | 66.3 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  |  |  |  | 2
  Male | 2 |  |  |  |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  |  |  | 0
  Asian | 0 |  |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  |  |  | 0
  Black or African American | 0 |  |  |  |  | 0
  White | 4 |  |  |  |  | 4
  More than one race | 0 |  |  |  |  | 0
  Unknown or Not Reported | 0 |  |  |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: This refers to the frequency of grade 3 or 4 AEs considered to be probably or definitely related to the treatment regimen. Toxicity will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE version [v] 5.0).
Time Frame: Up to 30 days post treatment initiation, On average, the timeframe is 25 days
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Participants | 0 |  |  |  |

2. Primary Outcome: Kinetics of Viral Load
Description: Will be assessed as cycle threshold values in nasopharyngeal swabs based on quantitative polymerase chain reaction (PCR) in the course of treatment and days 1, 3/4, 7, and 11.
Time Frame: Treatment and days 1, 3/4, 7 and 11
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Viral Copy Number / mL
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Viral Copy Number / mL
  C1D1 | 4300100.7 (5.9) |  |  |  |
  C1D3/4: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  C1D3/4 | 190808.2 |  |  |  |
  C1D7: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  C1D7 | 1974796.7 |  |  |  |
  C1D11: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  C1D11 | 16.6 |  |  |  |

3. Secondary Outcome: Number of Participants With Selected Clinical Efficacy Complications
Description: Will be assessed by the frequency of these complications: (i) progression of infection requiring hospitalization; (ii) respiratory failure requiring mechanical ventilation (primary efficacy endpoint); and (iii) death within 30 days. If present, acute respiratory distress syndrome will be graded by Berlin criteria.
Time Frame: Up to 30 days post treatment initiation
Population: All treated and evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Participants
  Total Number of Participants with complications | 2 |  |  |  |
  Number of participants that experienced progression of infection requiring hospitalization | 2 |  |  |  |
  Number of participants experienced failure requiring mechanical ventilation | 1 |  |  |  |
  Number of participants that died within 30 days | 2 |  |  |  |

4. Secondary Outcome: Kinetics of Viral Load
Description: Will be assessed as cycle threshold values in the peripheral blood and nasopharyngeal swab based on quantitative PCR in the course of treatment and days 1, 3, 7, and 14.
  Data entered are values that were measured, no "placeholders" were entered, zero is a valid measurement.
Time Frame: Days 1, 3, 7, 14 post treatment initiation
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
Relative mRNA abundance
  C1D1 | 0.0 (0.0) |  |  |  |
  C1D3: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  C1D3 | 0.0 |  |  |  |
  C1D7: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  C1D7 | 0.31 (0.43) |  |  |  |
  C1D14: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  C1D14 | 0.0 |  |  |  |

5. Secondary Outcome: Kinetics of Changes of the Immune Subsets and Circulating Inflammatory Mediators in Peripheral Blood (COX2)
Description: Gene expresssion measured by qPCR
Time Frame: Days 1, 4 , 7, 14 and 30 post treatment initiation
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.82 (0.65) |  |  |  |
  D1 Post | 0.68 (0.77) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 1.14 (0.99) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 1.0 (0.35) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 4.68 (6.92) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 1.67 (1.99) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 4.71 |  |  |  |

6. Secondary Outcome: Kinetics of Changes of the Immune Subsets and Circulating Inflammatory Mediators in Peripheral Blood (CCL5)
Description: Gene expression measured by QPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 23.0 (37.5) |  |  |  |
  D1 Post | 18.6 (30.5) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 32.0 (39.6) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 28.9 (17.0) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 19.6 (28.0) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 57.9 (60.0) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 116.7 |  |  |  |

7. Secondary Outcome: Kinetics of Changes of the Immune Subsets and Circulating Inflammatory Mediators in Peripheral Blood (CXCL10)
Description: Gene expression measured by qPCR
Time Frame: Days 1, 4, 7, 14, and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.01 (0.01) |  |  |  |
  D1 Post | 0.01 (0.01) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 0.03 (0.01) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.04 (0.01) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 0.04 (0.04) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 0.03 (0.002) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 0.05 |  |  |  |

8. Secondary Outcome: Kinetics of Changes of the Immune Subsets and Circulating Inflammatory Mediators in Peripheral Blood (CCL22)
Description: Gene expression measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.0013 (0.0007) |  |  |  |
  D1 Post: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D1 Post | 0.0001 (0.0001) |  |  |  |
  D4 Pre: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D4 Pre | 0.0023 |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.0018 (0.0013) |  |  |  |
  D7: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D7 | 0.0011 (0.0009) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 0.0043 (0.0050) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 0.0033 |  |  |  |

9. Secondary Outcome: Kinetics of Changes of the Immune Subsets and Circulating Inflammatory Mediators in Peripheral Blood (CXCL12)
Description: Gene expression measured by qPCR
Time Frame: Days 1, 4, 7, and 30 post treatment
Population: All treated and eligible patients, participants with data collected at each time point were analyzed.
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D1 Pre | 0.0038 (0.0006) |  |  |  |
  D1 Post: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D1 Post | 2,003.9 (3,470.8) |  |  |  |
  D4 Pre: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D4 Pre | 0.00021 |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.0011 (0.0012) |  |  |  |
  D7: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D7 | 0.0005 (0.0003) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 0.0039 |  |  |  |

10. Secondary Outcome: Kinetics of Changes of the Immune Subsets and Circulating Inflammatory Mediators in Peripheral Blood (IL-10)
Description: gene expression measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.075 (0.069) |  |  |  |
  D1 Post | 0.055 (0.064) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 0.059 (0.054) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.047 (0.033) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 0.072 (0.071) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 0.021 (0.007) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 0.014 |  |  |  |

11. Secondary Outcome: Kinetics of Changes of the Immune Subsets and Circulating Inflammatory Mediators in Peripheral Blood (IDO1)
Description: Gene expression measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Median (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.005 (0.008) |  |  |  |
  D1 Post | 0.007 (0.009) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 0.018 (0.00001) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.015 (0.003) |  |  |  |
  D7: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D7 | 0.019 (0.010) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 0.019 (0.010) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 0.029 |  |  |  |

12. Secondary Outcome: Kinetics of Changes of the Immune Subsets and Circulating Inflammatory Mediators in Peripheral Blood (IFNB1)
Description: Gene expression measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.19 (0.18) |  |  |  |
  D1 Post | 0.35 (0.48) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 0.83 (0.96) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.85 (1.03) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 0.50 (0.50) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 1.30 (1.56) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 1.68 |  |  |  |

13. Secondary Outcome: Kinetics of Changes of the Immune Subsets and Circulating Inflammatory Mediators in Peripheral Blood (IFNa)
Description: Gene expression measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.13 (0.12) |  |  |  |
  D1 Post | 0.22 (0.27) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 0.60 (0.65) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.68 (0.83) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 0.42 (0.42) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 0.82 (0.94) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 1.58 |  |  |  |

14. Secondary Outcome: Known Mediators of Antiviral Immunity (RIG-1)
Description: Induction of known mediator RIG-1 of antiviral immunity measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.27 (0.22) |  |  |  |
  D1 Post | 0.47 (0.42) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 0.50 (0.17) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.63 (0.30) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 0.45 (0.36) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 0.53 (0.33) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 1.16 |  |  |  |

15. Secondary Outcome: Known Mediators of Antiviral Immunity (TLR-3)
Description: Induction of known mediator TLR-3 of antiviral immunity measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.01 (0.01) |  |  |  |
  D1 Post | 0.02 (0.02) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 0.02 (0.03) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.03 (0.03) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 0.01 (0.01) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 0.04 (0.04) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 0.06 |  |  |  |

16. Secondary Outcome: Known Mediators of Antiviral Immunity (ISG-15)
Description: Induction of known mediator ISG-15 of antiviral immunity measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 1.29 (2.26) |  |  |  |
  D1 Post | 1.49 (2.62) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 0.02 (0.02) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.24 (0.02) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 0.37 (0.14) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 0.02 (0.002) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 0.23 |  |  |  |

17. Secondary Outcome: Known Mediators of Antiviral Immunity (RNAseL)
Description: Induction of known mediator RNAseL of antiviral immunity measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.06 (0.04) |  |  |  |
  D1 Post | 0.10 (0.06) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 0.10 (0.07) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.15 (0.07) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 0.13 (0.08) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 0.10 (0.08) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 0.28 |  |  |  |

18. Secondary Outcome: Known Mediators of Antiviral Immunity (OAS2)
Description: Induction of known mediator OAS2 of antiviral immunity measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 1.62 (1.44) |  |  |  |
  D1 Post | 1.92 (1.79) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 1.54 (0.82) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 2.94 (1.02) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 1.98 (1.30) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 2.30 (0.66) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 2.74 |  |  |  |

19. Secondary Outcome: Known Mediators of Antiviral Immunity (ACE2)
Description: Induction of known mediator ACE2 of antiviral immunity measured by qPCR
Time Frame: Days 1, and 14 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Post | 0.00012 (0.00013) |  |  |  |
  D14: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D14 | 0.0004 |  |  |  |

20. Secondary Outcome: Known Mediators of Antiviral Immunity (Mx1)
Description: Induction of known mediator Mx1 of antiviral immunity measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 2.42 (1.69) |  |  |  |
  D1 Post | 3.15 (2.81) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 2.60 (1.65) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 3.88 (1.57) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 3.13 (1.12) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 2.42 (1.12) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 3.40 |  |  |  |

21. Secondary Outcome: Known Mediators of Antiviral Immunity (IFIT1)
Description: Induction of known mediator IFIT1 of antiviral immunity measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.99 (0.56) |  |  |  |
  D1 Post | 1.29 (1.20) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 1.44 (1.34) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 2.14 (2.15) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 1.34 (1.00) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 2.22 (2.37) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 3.83 |  |  |  |

22. Secondary Outcome: Known Mediators of Antiviral Immunity (IFITM3)
Description: Induction of known mediator IFITM3 of antiviral immunity measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 17.45 (21.64) |  |  |  |
  D1 Post | 13.97 (13.93) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 11.10 (1.77) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 14.55 (1.07) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 12.48 (4.78) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 7.11 (0.96) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 5.93 |  |  |  |

23. Secondary Outcome: Known Mediators of Antiviral Immunity (IRF3)
Description: Induction of known mediator IRF3 of antiviral immunity measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 2.89 (2.83) |  |  |  |
  D1 Post | 3.04 (2.49) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 3.07 (3.33) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 4.14 (4.13) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 2.23 (2.08) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 4.26 (4.31) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 8.14 |  |  |  |

24. Secondary Outcome: Known Mediators of Antiviral Immunity (IRF7)
Description: Induction of known mediator IRF7 of antiviral immunity measured by qPCR
Time Frame: Days 1, 4, 7, 14 and 30 post treatment
Population: All treated and eligible patients
Measure: Mean (Standard Deviation); unit: Relative mRNA abundance
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 4 | 0 | 0 | 0 | 0
Relative mRNA abundance
  D1 Pre | 0.79 (8.88) |  |  |  |
  D1 Post | 0.41 (0.51) |  |  |  |
  D4 Pre: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Pre | 0.47 (0.45) |  |  |  |
  D4 Post: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D4 Post | 0.79 (0.58) |  |  |  |
  D7: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  D7 | 0.54 (0.47) |  |  |  |
  D14: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0
  D14 | 0.49 (0.40) |  |  |  |
  D30: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
  D30 | 0.91 |  |  |  |

25. Other Pre Specified Outcome: Known Mediators of Antiviral Immunity
Description: Will assess the induction of known mediators of antiviral immunity that include (myxovirus resistance gene, MxA; protein Kinase R; oligoadenylate synthetase-2; RNAse-L, IFN-stimulated gene-15 (ISG15); IFN-induced proteins with tetratricopeptide repeats, and IFN-inducible transmembrane protein 3, TLR3, RIG-I, MDA5, IRF3, IRF7, in nasopharyngeal swabs material and blood cells of patients on all tiers of treatment. Will also assess the expression of ACE2 (receptor for severe acute respiratory syndrome coronavirus 2 [SARS-Cov-2] entry) and potentially other genes involved in SARS-CoV-2 infection will be tested in nasopharyngeal samples.
Time Frame: Up to 30 days post treatment initiation
Population: No patients were evaluable.
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Routine AEs occurring between the start date of intervention until 30 days after the last intervention, or until the event has resolved, the study participant is lost to follow-up, the start of a new treatment, or until the study investigator assesses the event(s) as stable or irreversible, will be reported. up to 30 days post treatment initiation for an average timeframe of 25 days.
Description: Due to the study's early termination, as a result of low accrual, target accrual was not reached, and additional treatment arms were not accrued.
Groups:
- 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2: "Dose level 2 :Patients receive rintatolimod IV over 2.5-3 hours plus recombinant interferon alfa-2b IV 5 MU/M^2 over 20 minutes on day 1 and on day 3 (or 4) in the absence of disease progression or unacceptable toxicity.
  Biological/Vaccine: Recombinant Interferon Alfa-2b Given IV
  Other Names:
  Alfatronol Glucoferon Heberon Alfa IFN alpha-2B Interferon alfa 2b Interferon Alfa-2B Interferon Alpha-2b Intron A recombinant interferon alfa-2b Sch 30500 Urifron Viraferon Drug: Rintatolimod Given IV
  Other Names:
  Ampligen Atvogen RINTATOLIMOD"
- 3. Experimental: Rrintatolimod Plus Standard of Care): "Patients receive rintatolimod IV over 2.5-3 hours once plus standard of care.
  Drug: Rintatolimod Given IV
  Other Names:
  Ampligen Atvogen RINTATOLIMOD"
- 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2: "Dose level 3: Patients receive rintatolimod IV over 2.5-3 hours plus recombinant interferon alfa-2b IV 10 MU/M^2 over 20 minutes on day 1 and on day 3 (or 4) in the absence of disease progression or unacceptable toxicity.
  Biological/Vaccine: Recombinant Interferon Alfa-2b Given IV
  Other Names:
  Alfatronol Glucoferon Heberon Alfa IFN alpha-2B Interferon alfa 2b Interferon Alfa-2B Interferon Alpha-2b Intron A recombinant interferon alfa-2b Sch 30500 Urifron Viraferon Drug: Rintatolimod Given IV
  Other Names:
  Ampligen Atvogen RINTATOLIMOD"
- 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2: "Dose level 4: Patients receive rintatolimod IV over 2.5-3 hours plus recombinant interferon alfa-2b IV 20 MU/M^2 over 20 minutes on day 1 and on day 3 (or 4) in the absence of disease progression or unacceptable toxicity.
  Biological/Vaccine: Recombinant Interferon Alfa-2b Given IV
  Other Names:
  Alfatronol Glucoferon Heberon Alfa IFN alpha-2B Interferon alfa 2b Interferon Alfa-2B Interferon Alpha-2b Intron A recombinant interferon alfa-2b Sch 30500 Urifron Viraferon Drug: Rintatolimod Given IV
  Other Names:
  Ampligen Atvogen RINTATOLIMOD"
Arm/Group | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 | 3. Experimental: Rrintatolimod Plus Standard of Care) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2
All-Cause Mortality (participants affected / at risk) | 3/4 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/4 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 (N=4) | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 (N=0) | 3. Experimental: Rrintatolimod Plus Standard of Care) (N=0) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 (N=0) | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2 (N=0)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | NA | NA | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 0 MU/M^2 (N=4) | 2. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 5 MU/M^2 (N=0) | 3. Experimental: Rrintatolimod Plus Standard of Care) (N=0) | 4. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 10 MU/M^2 (N=0) | 5. Experimental: Rintatolimod, Recombinant Interferon Alfa-2b 20 MU/M^2 (N=0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | NA | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | NA | NA | NA | NA
Diarrhea (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 1 (1) | NA | NA | NA | NA
Edema limbs (General disorders) | 1 (1) | NA | NA | NA | NA
Fatigue (General disorders) | 2 (2) | NA | NA | NA | NA
Flu like symptoms (General disorders) | 1 (1) | NA | NA | NA | NA
Sinusitis (Infections and infestations) | 1 (1) | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 1 (1) | NA | NA | NA | NA
Platelet count decreased (Investigations) | 1 (1) | NA | NA | NA | NA
Depression (Psychiatric disorders) | 1 (1) | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 1 (1) | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA | NA | NA
Hypotension (Vascular disorders) | 1 (1) | NA | NA | NA | NA
Thromboembolic event (Vascular disorders) | 1 (1) | NA | NA | NA | NA

LIMITATIONS AND CAVEATS:
Due to the study's early termination, as a result of low accrual, target accrual was not reached and no statistical inference of the primary and secondary aims were carried forth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT04379518/Prot_SAP_000.pdf